CLINICAL TRIAL: NCT06262568
Title: Effect of Instructional Guidelines on Maternity Nurses' Awareness Toward High Risk Pregnancy and Maternal Near Miss Cases
Brief Title: Effect of Guidelines on Nurses' Awareness Toward HRP and Maternal Near Miss Cases
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Hazem Mohamed, Clinical demonstrator, Obstetrics and Gynecology Nursing- Faculty of Nursing, Sohag University, Sohag University
Other Study IDs: Soh-Med-23-03-18MS
Record Dates: First submitted 2023-12-20; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: High Risk Pregnancy and Maternal Near Miss Cases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assess the nurse knowledge and practices. — assess the nurse knowledge and practices.

SUMMARY:
The current study will evaluate the impact of awareness of maternity nurses toward instructional guidelines and evaluate the knowledge, practice and attitude of nurses toward high risk pregnancy and maternal near miss cases before and after education.

DETAILED DESCRIPTION:
Maternal morbidity is defined as ill-health in a woman during pregnancy, irrespective of pregnancy site or duration, which is caused or aggravated by the pregnancy or its management, but which is not caused by accident or incident. This concept ranges from mild to severe maternal morbidity (SMM). Maternal near-miss (MNM) and potentially life-threatening conditions (PLTCs) are included as SMM.(Mekonnen et al., 2021) . Maternal mortality is an indicator of many parameters of maternal health, such as women's status, access to care and quality of care in low resource settings.(Mohammed et al., 2020) Maternal near-miss precedes maternal mortality, and women are still alive indicating that the numbers of near-misses occur more often than maternal mortality.(Mekonnen et al., 2021) Maternal near miss case is defined as "a woman who nearly died but survived a complication that occurred during pregnancy, childbirth, or within 42 days of termination of pregnancy"(Ninama et al., 2022) High risk pregnancy is defined as one where pregnancy is complicated by factor or factors that adversely affects the outcome- maternal or perinatal or both. Women with high-risk pregnancies should receive care from a special team of health care providers to ensure the best possible outcomes. (Arjariya & Tiwari, .2021) .High-risk pregnancy was classified based on the guidelines provided by Pradhan Mantri Surakshit Matritva Abhiyan (PMSMA) for identification of high-risk pregnancy by health-care workers. The parameters considered for diagnosis of high- risk pregnancy were also defined as per the guidelines provided by PMSMA. Antenatal women with the following conditions were categorized under high-risk pregnancy: a. Severe anemia with hemoglobin level 140/90 mmHg) b. Hypertensive disorder in pregnancy (blood pressure >140/90 mmHg) c. Previous history of lower segment cesarean section d. Bad obstetric history (history of obstructed labor) e. Low-lying placenta or placenta previa. .(Arjariya & Tiwari.,2021)

ELIGIBILITY:
Inclusion Criteria:

* all nurses staff

Exclusion Criteria:

* nurses who refuse participation

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: all nurses
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the outcome of instructional guidelines on maternity nurses' awareness toward high-risk pregnancy and Maternal Near Miss Cases by questionnaire before and after training | 10 months
  Evaluate the outcome of instructional guidelines on maternity nurses' awareness toward high-risk pregnancy and Maternal Near Miss Cases by questionnaire before and after training

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided